CLINICAL TRIAL: NCT02621333
Title: Chemotherapy Combined Autologous Cytokine-induced Killer Cells in Naive Stage IV EGFR-wild Type Lung Adenocarcinoma: A Prospective, Randomised, Open, Multicenter Phase Ⅱ Study
Brief Title: Chemotherapy Combined Autologous Cytokine-induced Killer Cells in Naive Stage IV EGFR-wild Type Lung Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: As there are so many clinical trials in progress and the number of patients enrolled limited.
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Henan Provincial People's Hospital (Other); Hebei Medical University Fourth Hospital (Other); Shanxi Dayi Hospital (Other); Tangshan People's Hospital (Other); 150th Hospital of PLA (Other Government); First Affiliated Hospital of Nanyang Medical College (Other); Nanyang Central Hospital (Other); First People's Hospital of Shangqiu (Other); Anyang Regional Hospital (Other); Puyang Oilfield General Hospital (Other); Shenma Medical Group General Hospital (Other); Jiaozuo Tumor Hospital (Unknown); The 152th Central Hospital of PLA (Other); Xinyang Central Hospital (Other)
Responsible Party: Principal Investigator, Quanli Gao, director, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HenanCH003
Record Dates: First submitted 2015-11-25; First posted 2015-12-03 (Estimated); Last update posted 2021-05-12 (Actual); Status verified 2020-02

CONDITIONS: Lung Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CIK combined chemotherapy group (Experimental): autologous CIK combined chemotherapy group Drugs: platinum combined doublets; After 3 or 4 days of chemotherapy, about 5×109 autologous cytokine-indued killer cells are transfused into the vein of patients in one hour.
  Interventions: Biological: CIK; Drug: chemotherapy
- chemotherapy group (Active Comparator): platinum combined doublets Drugs: Paclitaxel 175mg/m2 D1, or Docetaxel75mg/m2 D1, or Pemetrexed Disodium 500mg/m2，D1；combined cisplatin 25mg/ m2，D1-3 or carboplatin AUC=5, D1.
  Interventions: Drug: chemotherapy

INTERVENTIONS:
Biological: CIK — platinum combined doublets: Paclitaxel 175mg/m2 D1, or Docetaxel75mg/m2 D1, or Pemetrexed Disodium 500mg/m2，D1；combined cisplatin 25mg/m2，D1-3 or carboplatin AUC=5, D1. After 3 or 4 days of chemotherapy, about 5×109 autologous cytokine-induced killer cells are transfused into the vein of patients in one hour.
  Other Names: autologous cytokine-induced killer cells
  Arms: CIK combined chemotherapy group
Drug: chemotherapy — platinum combined doublets: Paclitaxel 175mg/m2 D1, or Docetaxel75mg/m2 D1, or Pemetrexed Disodium 500mg/m2，D1；combined cisplatin 25mg/m2，D1-3 or carboplatin AUC=5, D1.
  Other Names: platinum combined doublets

SUMMARY:
This is a prospective, randomized, open, multicenter phase Ⅱ study to evaluate the efficacy of cytokine-induced killer cells combined chemotherapy in stage Ⅳ naive EGFR wild-type lung adenocarcinoma.

DETAILED DESCRIPTION:
There is still no great improvement in advanced EGFR wild-type lung adenocarcinoma although great progress was made in treatment of non-small cell lung cancer. It's necessary to explore the treatment mode of this kind of patients. As the progress was made in tumor immunity and immunotherapy, more and more cancer therapists accept the treatment model of chemotherapy combined immunotherapy. And now chemotherapy combined autologous CIK cells is one kind of common treatment model in some countries. Investigators try to evaluate the efficacy and safety of this kind of treatment model in patients with stage Ⅳ naive EGFR wild-type lung adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as stage Ⅳ naive EGFR wild-type lung adenocarcinoma by image, tissue and/or cytology; or relapse after operation (if the patient received adjuvant chemotherapy and the interval between the last chemotherapy and relapse is at least six months. The detection method of EGFR mutation is ARMS.
2. EML4-ALK fuse gene is negative and the detection of EML4-ALK is FISH or ventana IHC.
3. There should be at least one measurable lesions (by CT or MRI)
4. No other cancer history ( except skin squamous cell carcinoma after surgery)
5. Age between 18 and 75 years old
6. World health organization- Eastern Cooperative Oncology Group Performance Status 0-1
7. Life expectancy more than 3 months and can be followed-up
8. Patients must have adequate organ and marrow functions as defined below: white blood cells: more than 3.5×109/L, Neutrophils: more than 1.5×109/L, Platelets: more than 80×109/L, Hemoglobin more than 90g/L, Serum total bilirubin less than 1.5 folds of the upper normal limit (ULN), Serum glutamic-oxal

   (o) acetic transaminase: less than 2.5×ULN (if there is liver metastasis less than 5×ULN); Serum creatinine: less than 1.0×ULN, Prothrombin time, Active partial thromboplastin time, Fibrinogen, Thrombin time are in normal ranges.
9. Women of child-bearing period must take effective contraceptive measures during all the time of study. During the period of study the results of blood and urine pregnancy test should be negative.
10. Men should take effective contraceptive measures from the beginning of therapy to one month after the last cycle of chemotherapy.
11. Willing to comply with the ban and constraints for this study protocol specified.
12. Informed consent and willing to participate in this study.

Exclusion Criteria:

1. Accepted other study drugs 30 days before the beginning of this study.
2. Brain metastases with clinical symptoms ( with exception of being controlled after radiation)
3. Active viral or bacterial infection and can't be controlled with appropriate anti-infection treatment
4. Known as HIV infection, syphilis serology reaction positive, active hepatitis B virus or hepatitis C virus infection
5. Suffering from mental illness or other illness, such as heart or lung disease, diabetes, etc. that can not be controlled, and can not be coped with study treatment and monitoring requirements.
6. Known allergy to any kind of component of study drugs
7. Active rheumatic diseases
8. Organ transplant recipients
9. Poor compliance
10. Pregnant women
11. Lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
overall survival time | from the day of randomization to the day of death, up to 36 months
  overall survival time aims at from date of randomization until the date of death from any cause, up to 36 months

SECONDARY OUTCOMES:
time to progression | from the day of randomization to the day of first detecting progression, up to 24 months
  time to progression points to from date of randomization until the date of first documented progression, up to 24 months
objective response rate | one year
  the partion of overall remission in total proportion

CONTACTS AND LOCATIONS:
Overall Officials: Quanli Gao, M.D., Study Director — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital/The affiliated Cancer Hospital of ZhengZhou university, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No
terminated as the slow enrollment

REFERENCES:
- [Result] Li R, Wang C, Liu L, Du C, Cao S, Yu J, Wang SE, Hao X, Ren X, Li H. Autologous cytokine-induced killer cell immunotherapy in lung cancer: a phase II clinical study. Cancer Immunol Immunother. 2012 Nov;61(11):2125-33. doi: 10.1007/s00262-012-1260-2. Epub 2012 May 13. PMID 22581306
- [Result] Zhong R, Teng J, Han B, Zhong H. Dendritic cells combining with cytokine-induced killer cells synergize chemotherapy in patients with late-stage non-small cell lung cancer. Cancer Immunol Immunother. 2011 Oct;60(10):1497-502. doi: 10.1007/s00262-011-1060-0. Epub 2011 Jun 17. PMID 21681372
- [Result] Wang S, Wang Z. Efficacy and safety of dendritic cells co-cultured with cytokine-induced killer cells immunotherapy for non-small-cell lung cancer. Int Immunopharmacol. 2015 Sep;28(1):22-8. doi: 10.1016/j.intimp.2015.05.021. Epub 2015 May 23. PMID 26013109
- [Derived] Zhao L, Li W, Wang Z, Yang Y, Zhang Y, Shang Y, Ren X, Gao Q. Survival benefit from RectroNectin-activated cytokine-induced killer cells combined with chemotherapy in advanced EGFR wild-type lung adenocarcinoma. Immunotherapy. 2018 Mar 1;10(6):501-510. doi: 10.2217/imt-2017-0140. PMID 29562855